CLINICAL TRIAL: NCT05986435
Title: Long-term Large Sample Multicenter Follow-up Study of COVID-19
Brief Title: Long-term Follow-up Study of COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Qin Ning, Director, department of infection, Tongji Hospital
Other Study IDs: PROCOVER
Record Dates: First submitted 2023-08-08; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — There are many patients who are prospectively observed. Their samples will be collected. The samples will include blood, urine, throat swabs etc.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn the long-term prognosis of patients and the clinical characteristics of complications, which is of great significance for treatment of novel coronavirus infection pneumonia.

This trial plans to include 5700 inpatients with positive SARS CoV-2 nucleic acid test results. This trial does not involve the use of specific drug. Participants's health and psychological status will be observed at the preset time points. The blood, feces, urine samples of patients will be collected for relevant tests.

DETAILED DESCRIPTION:
After the patients are enrolled, record the patient's treatment regimens, blood routine results, blood biochemistry results, cytokines results, lung imaging results, and cranial imaging results, understand the patient's current clinical manifestations, evaluate the patient's psychological status and quality of life, and collect samples of the patients' blood, feces, urine, and other related tests.

Collection of clinical samples: collect blood, urine, throat swabs and other samples from patients with confirmed novel coronavirus pneumonia (Nucleic acid test positive), and collect samples for relevant tests at 3 months, 6 months, 12 months, 18 months, 24 months and 36 months after discharge of patients, and record the clinical manifestations of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed COVID-19

Exclusion Criteria:

* Combined infection with influenza virus, mycoplasma, and chlamydia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The inpatients with positive SARS CoV-2 nucleic acid test results will be included.
Sampling Method: Probability Sample
Enrollment: 5700 (Estimated)
Dates: Start 2020-10-20 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
clinical manifestation | 3 months, 6 months, 12 months, 18 months, 24 months, 36 months after patients discharge

SECONDARY OUTCOMES:
psychological status | 3 months, 6 months, 12 months, 18 months, 24 months, 36 months after patients discharge
quality of life scores | 3 months, 6 months, 12 months, 18 months, 24 months, 36 months after patients discharge
cranial imaging results | 3 months, 6 months, 12 months, 18 months, 24 months, 36 months after patients discharge
lung imaging results | 3 months, 6 months, 12 months, 18 months, 24 months, 36 months after patients discharge
cytokines level | 3 months, 6 months, 12 months, 18 months, 24 months, 36 months after patients discharge
blood biochemistry results | 3 months, 6 months, 12 months, 18 months, 24 months, 36 months after patients discharge
routine blood test results | 3 months, 6 months, 12 months, 18 months, 24 months, 36 months after patients discharge
treatment regimens | 3 months, 6 months, 12 months, 18 months, 24 months, 36 months after patients discharge
survival rate | 3 months, 6 months, 12 months, 18 months, 24 months, 36 months after patients discharge

CONTACTS AND LOCATIONS:
Overall Officials: Qin Ning, Professor, Principal Investigator — Tongji Hospital
Locations (2):
- China (2):
  - Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science & Technology, Wuhan, Hubei
  - Wuhan Seventh Hospital, Wuhan, Hubei